CLINICAL TRIAL: NCT03662698
Title: Effect of Guided Imagery for Radiotherapy-Related Distress: A Randomized, Controlled Trial for Patients With Head and Neck Cancer
Brief Title: Effect of Guided Imagery for Radiotherapy-Related Distress in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18-1100.cc
Record Dates: First submitted 2018-08-31; First posted 2018-09-07 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cancer
Keywords: Radiotherapy; Guided Imagery; Therapy; Distress; Anxiety; Depression
MeSH Terms: conditions — Head and Neck Neoplasms; Anxiety Disorders; Depression | interventions — Imagery, Psychotherapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the guided imagery intervention or to treatment as usual.
Who Masked: Outcomes Assessor
Masking Description: Due to study design, it is not possible to blind either participants or investigators to study condition. However, the biostatistician will be blinded to participant group to minimize bias in analyzing the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Imagery (Experimental): The GI intervention will include direct, written, and audio delivery of one of three GI vignettes (depiction).The patient will be able to choose one of the three vignettes.
  Interventions: Behavioral: Guided Imagery
- Treatment as Usual (Active Comparator): The control, or treatment as usual condition, will include an orientation to radiotherapy from the clinic nurse coordinator.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Guided Imagery — GI is a relaxation technique involving the visualization of images and is considered an adjuvant cancer therapy.The GI intervention will include two hour-long meetings between the participant and a trained interventionist. The sessions will include direct, written, and audio delivery of one of three GI vignettes. The patient will be able to choose one of the three vignettes. The approximately twelve minute long vignettes included in the study will be: Taking a Walk, Healthy Cell Alliance for Treatment, and Daily Intention (32). Patients will also be given access to psychosocial support resources (i.e., clinical psychologists and social workers) at University of Colorado Cancer Center.
  Arms: Guided Imagery
Other: Treatment as Usual — This will include a tour of the treatment room and education about RT. Patients will also receive educational materials about RT including the process of RT and CT simulation, treatment side effects, pain management, and swallowing exercises. Participants in this condition will also have access to psychosocial support resources (i.e., clinical psychologists and social workers) at University of Colorado Cancer Center.
  Arms: Treatment as Usual

SUMMARY:
The goal of this interdisciplinary pilot study is to evaluate the feasibility, acceptability and preliminary efficacy of a guided imagery intervention to reduce radiotherapy-related symptoms of anxiety and depression in patients with head and neck cancers relative to treatment as usual.

DETAILED DESCRIPTION:
The goal of this interdisciplinary pilot study is to evaluate the feasibility, acceptability and preliminary efficacy of a guided imagery intervention to reduce radiotherapy-related symptoms of anxiety and depression in patients with head and neck cancers relative to treatment as usual. Treatment as usual contains no psychological interventions to aid in distress, however participants will have access to the psychosocial supports at the cancer center available to all patients. Patients will be randomized to either condition, and surveys of their well-being will be conducted throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be aged 18 - 100.
4. Ability to read and communicate in English.
5. A confirmed malignancy of the head and neck region (including metastases from other primary tumors and cancers of unknown primary.
6. Initiation of RT at the University of Colorado Cancer Center.
7. Psychiatric and cognitive stability as assessed by chart review (i.e., no documented dementia diagnosis or unmanaged psychiatric symptoms) and study personnel (i.e., ability to attend to meeting with study personnel).
8. Ability to meet remotely via internet connection or over the phone.

Exclusion Criteria:

1. Any individual who does not meet the inclusion criteria.
2. Those who are determined, by mental health professionals, to be psychiatrically unstable.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Kolva, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Derived] Kolva E, Karam SD, Carr AL, Roberts S, Torkko K, Lanning R, Cox-Martin E. Guided imagery for treatment (GIFT): protocol of a pilot trial of guided imagery versus treatment as usual to address radiotherapy-related distress in head and neck cancer. Pilot Feasibility Stud. 2022 Sep 5;8(1):199. doi: 10.1186/s40814-022-01134-9. PMID 36064748

RESULTS

PARTICIPANT FLOW:
Groups:
- Guided Imagery: The GI intervention will include direct, written, and audio delivery of one of three GI vignettes (depiction).The patient will be able to choose one of the three vignettes.
  Guided Imagery: GI is a relaxation technique involving the visualization of images and is considered an adjuvant cancer therapy.The GI intervention will include two hour-long meetings between the participant and a trained interventionist. The sessions will include direct, written, and audio delivery of one of three GI vignettes. The patient will be able to choose one of the three vignettes. The approximately twelve minute long vignettes included in the study will be: Taking a Walk, Healthy Cell Alliance for Treatment, and Daily Intention (32). Patients will also be given access to psychosocial support resources (i.e., clinical psychologists and social workers) at UCCC.
- Treatment as Usual: The control, or treatment as usual condition, will include an orientation to RT from the clinic nurse coordinator.
  Treatment as Usual: This will include a tour of the treatment room and education about RT. Patients will also receive educational materials about RT including the process of RT and CT simulation, treatment side effects, pain management, and swallowing exercises. Participants in this condition will also have access to psychosocial support resources (i.e., clinical psychologists and social workers) at UCCC.
Period: Overall Study
Arm/Group | Guided Imagery | Treatment as Usual
Started | 26 | 31
Completed | 19 | 25
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guided Imagery | Treatment as Usual | Total
Number analyzed (Participants) | 26 | 31 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 6 | 12 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (14.3) | 62.6 (9.6) | 60.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 18 | 26 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 24 | 29 | 53
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 31 | 57

OUTCOME MEASURES:

1. Primary Outcome: The Desire for Patients to Want to Use Guided Imagery While Undergoing Radiotherapy: [Feasibility]
Description: Feasibility of intervention use will be assessed through rates of study completion.
Time Frame: From baseline to one month post-radiotherapy.
Population: A total of 192 or 373 (51%) of radiation oncology patients were eligible based on pre-screening criteria. 125 were approached and 57 (45.6%) consented for participation. Most participants (n= 44, 77.2%) completed participation in the study. One participant withdrew due to treatment plan changes, the others did not provide reasons, or were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Guided Imagery | Treatment as Usual
Number analyzed (Participants) | 26 | 31
Participants | 19 | 25

2. Primary Outcome: The Desire for Patients to Want to Use Guided Imagery While Undergoing Radiotherapy: [Feasibility]
Description: Feasibility of intervention use will be assessed through rates of GI session attendance.
Time Frame: From baseline to week one of radiotherapy.
Population: 21 participants were scheduled for guided imagery sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Guided Imagery
Number analyzed (Participants) | 21
Participants
  Participants who completed two sessions of guided imagery | 18
  Participants who completed one session of guided imagery | 3

3. Primary Outcome: The Desire for Patients to Want to Use Guided Imagery While Undergoing Radiotherapy: [Feasibility]
Description: Feasibility of intervention use will be assessed through self-reported use of the GI intervention measured through timeline follow-back.
Time Frame: From baseline to one month post-radiotherapy, up to 12 weeks.
Population: Participants in the guided imagery arm reported on weekly use of the guided imagery intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Guided Imagery
Number analyzed (Participants) | 26
Participants
  Participants who used intervention at time of CT simulation | 4
  Participants who used intervention at week one | 10
  Participants who used intervention at week two | 9
  Participants who used intervention at week three | 11
  Participants who used intervention at week four | 13
  Participants who used intervention at week five | 9
  Participants who used intervention at week six | 9
  Participants who used intervention at week seven | 6
  Participants who used intervention at week twelve | 0

4. Primary Outcome: The Amount of Patients Who Find Using Guided Imagery Beneficial as a Form of Treatment While Undergoing Radiotherapy: [Acceptability]
Description: Acceptability of the intervention will be assessed through qualitative interviews with intervention participants. The interviews will assess participant experience in the intervention including thoughts about the intervention content and structure of the intervention. Qualitative data regarding acceptability of the intervention will be gathered through one-on-one, standardized open-ended interviews.
Time Frame: From baseline to one month post-radiotherapy.
Population: Participants in the guided imagery arm who completed the study participated in a qualitative interview about their experience. Data were assessed qualitatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Guided Imagery
Number analyzed (Participants) | 19
Participants
  Participants completed survey: Yes | 19
  Participants completed survey: No | 0
  Intervention was beneficial to participant: Yes | 17
  Intervention was beneficial to participant: No | 2

5. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scales (HADS) Score
Description: Assess the impact of the GI intervention on symptoms of anxiety and depression in patients with head and neck cancer using the Hospital Anxiety and Depression Scale (HADS).
  HADS is a 14-item self-report measure of anxiety and depression symptoms for use in a medically-ill patients. The measure contains 7 anxiety items and 7 depression items, corresponding to the two subscales. Each item is assessed with a 4 point Likert scale (range: 0-3) and the participant is asked to identify how much a given statement is applicable (Most of the time, A lot of the time, From time to time, Occasionally or Not at all). Subscale scores range from 0 to 21 with higher scores indicating greater severity of symptoms. A score of 8 on either subscale identifies cases of anxiety or depressive disorders.
  The total score is reported here, which is summed from the subscale scores. Min = 0, Max = 42.
Time Frame: Baseline and completion of radiotherapy at 7 weeks
Population: Patients were compared to themselves as well as across groups. We reviewed difference from screening to week 7. Some patients did not complete the assessment at week 7.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guided Imagery | Treatment as Usual
Number analyzed (Participants) | 14 | 21
units on a scale | 1.93 (8.95) | -0.05 (4.76)

6. Secondary Outcome: Change From Baseline in Memorial Symptom Assessment Scale Short Form (MSAS-SF) Score
Description: Assess the impact of the GI intervention on symptoms of anxiety and depression in patients with head and neck cancer using the Memorial Symptom Assessment Scale Short Form (MSAS-SF). The MSAS-SF assesses the occurrence of 26 physical symptoms and four psychological symptoms from 0 ("no symptom"), rarely (1), occasionally (2), frequently (3), and almost constantly (4). The distress that each symptom causes to the respondent is rated on a 5-point scale (again with range 0-4) including "not at all", "a little bit", "somewhat", "quite a bit", and "very much". Responses regarding symptom distress are used to create the Total Symptom Distress score (TMSAS), which is the average of the symptom scores across all symptoms in the form. The minimum value is 0 and the maximum value is 4. Higher scores indicate that the patient experienced a greater level of distress, which is a worse outcome. What is reported is the difference in score from baseline.
Time Frame: Baseline and end of radiotherapy at 7 weeks.
Population: Patients were compared to themselves as well as across groups. We reviewed difference from screening to 7 weeks. Some patients did not complete the assessment at week 7.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guided Imagery | Treatment as Usual
Number analyzed (Participants) | 13 | 19
units on a scale | -0.08 (0.64) | -0.11 (0.46)

7. Secondary Outcome: The Effect Guided Imagery Has on Distress While Undergoing Radiotherapy: [Impact]
Description: Assess the impact of the GI intervention on symptoms of anxiety and depression in patients with head and neck cancer using the Functional Assessment of Cancer Therapy-Head and Neck Version (FACT-HN). The FACT-HN is a 27-item self-report instrument designed to assess quality of life for patients with head and neck cancer. Items assess four domains: physical, social/family, emotional, and functional well-being (scores ranging 0 to 28) as well as specific items assessing head and neck symptoms. The scale uses a Likert-type scale (0 to 4) to produce subscale and total scores (ranging from 0-108) with higher scores indicating higher quality of life. It is a reliable, valid measure of quality of life for patients with head and neck cancer.
Time Frame: From baseline to completion of radiotherapy at 7 weeks.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guided Imagery | Treatment as Usual
Number analyzed (Participants) | 13 | 21
units on a scale | -16.54 (21.05) | -14.9 (21.2)

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Guided Imagery | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/31
Other Adverse Events (participants affected / at risk) | 0/26 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guided Imagery (N=26) | Treatment as Usual (N=31)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT03662698/Prot_SAP_000.pdf